CLINICAL TRIAL: NCT02059382
Title: EXercise Continuation Incorporating Technology Enhancements (EXCITE) Study
Acronym: EXCITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-10688
Record Dates: First submitted 2013-12-24; First posted 2014-02-11 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Physical Inactivity
Keywords: daily physical activity; exercise; social support; online social network
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): ChiRunning training Weekly training log Blinded accelerometer
  Interventions: Behavioral: ChiRunning training
- Technology support for behavior change (Experimental): ChiRunning training unblinded accelerometer tracking structured exercise using mobile app participation in online social network participation in study website
  Interventions: Behavioral: ChiRunning training; Behavioral: unblinded accelerometer; Behavioral: participation in online social network; Behavioral: participation in study website; Behavioral: Technology support for behavior change

INTERVENTIONS:
Behavioral: ChiRunning training
Behavioral: unblinded accelerometer
  Arms: Technology support for behavior change
Behavioral: participation in online social network
  Arms: Technology support for behavior change
Behavioral: participation in study website
  Arms: Technology support for behavior change
Behavioral: Technology support for behavior change
  Arms: Technology support for behavior change

SUMMARY:
The purpose of this study is to inform the integration of mobile and social media components into larger interventions aimed at increasing adherence and maintenance of physical activity. Nearly half of the US population do not meet physical activity recommendations of ≥150 minutes of moderate activity per week. The use of smartphones to "self track" data and upload that data to an online social network is becoming increasingly common and may be an effective way to motivate physical activity adherence and maintenance. We are proposing a two phase study to develop and evaluate a mobile health ("mHealth") intervention that includes the use of two existing technologies: 1) the RunKeeper mobile app to collect and upload exercise data (distance, pace, time), and 2) the RunKeeper.com online social network as a place to analyze uploaded data and engage with a coach and online community. Phase 1 (n=10) will iteratively develop the mHealth intervention and phase 2 (n=30) will pilot the mHealth intervention (participants will be randomized to either mHealth intervention (n=20) or control (n=10)) to collect feasibility, acceptability and preliminary efficacy data. All participants will attend a day-long ChiWalk/Run training to help them avoid potential injuries and meet their coach and community in-person. All participants will also be asked to wear a FitBit accelerometer from one week before the beginning of the intervention through one week after the end of the intervention to collect total physical activity data. This data will be uploaded automatically to the study data base. Primary outcomes will be total physical activity as collected by the FitBit accelerometer (and the RunKeeper mobile app for the intervention group) and secondary outcomes will be changes in psychological factors that may mediate adherence to physical activity.

ELIGIBILITY:
Inclusion Criteria:

* healthy underactive adults interested in using mobile and web based technologies to increase their physical activity
* low risk of cardiovascular disease
* comfortable reading and communicating in English
* owns a smartphone and is does not regularly use a fitness tracking mobile app
* has regular access to the internet and a wireless connection for data uploading.

Exclusion Criteria:

* currently meeting/exceeding recommend 450 MET min per week
* previous condition that would contraindicate regular moderate to vigorous physical activity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | End of 8 weeks of recruitment
  Meeting 75% of recruitment goal of 40 participants
Feasibility of retention | End of 10 weeks of participation
  Retaining 75% of enrolled participants.
Feasibility for participant adherence | Measured through out the 10 weeks of active participation
  Whether participants complete at least 75% of the exercise that they committed to at the beginning of the study.
Acceptability of study procedures | End of 10 weeks of active participation
  Did participants find study procedures acceptable?

SECONDARY OUTCOMES:
Total number of new exercise related injury | Measured through out the 10 weeks of active participation
  Measure of pain or injury associated with structured exercise.
Average weekly physical activity in steps | Measured through out the 10 weeks of active participation
  Daily step measured using a digital accelerometer.
Average weekly MET min of structured exercise | Measured through out the 10 weeks of active participation
  Average weekly metabolic equivalent of task (MET) minutes are a measure of time and intensity of physical activity.
Change in mindfulness | Baseline and end of 10 weeks of active participation
  We will use the Five Factor Mindfulness Questionnaire (FFMQ) to assess changes in mindfulness. FFMQ is a 39-item questionnaire with five subscales (observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience) and a summary score ranging from 39 to 195. Internal consistencies range from α=0.75-0.91.
Change in body awareness | Baseline and end of 10 weeks of active participation
  We used the Multi-dimensional Assessment of Interoceptive Awareness (MAIA) to measure body awareness. MAIA is a 32-item questionnaire with eight separately scored scales. .We used 3 of the 8 scales most relevant for an exercise intervention to assess body awareness. The subscales we used were: 1) Self-Regulation: ability to regulate distress by attention to body sensations; 2) Body Listening: active listening to the body for insight; 3) Trusting: experience of one's body as safe and trustworthy. Scales range from 0-5 with higher numbers representing higher aspects of body awareness with internal consistencies of α=0.83; 0.82; 0.79 on the Self-Regulation, Body Listening, and Trusting subscales, respectively.
Change in exercise self efficacy | Baseline and end of 10 weeks of active participation
  We will be using Multidimensional Self-Efficacy for Exercise Scale (MSES) to assess exercise related self efficacy. MSES is a 9-item instrument used to assess three dimension of exercise related self efficacy (task, scheduling and coping).
Change in social support | Baseline and end of 10 weeks of active participation
  We will use the Social support and exercise survey (SSES) to assess social support. SSES is 26 item survey of social support for exercise available to the individual using separate (13 item) scales each for friends and for family.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly McDermott, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States